CLINICAL TRIAL: NCT06886555
Title: Impact of Timing of Neuraxial Analgesia on Obstetric, Anesthesiologic and Neonatal Outcomes in Induced Labour
Acronym: TAIL
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Silvia Poma, Medical doctor- Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: TAIL
Record Dates: First submitted 2025-02-25; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Labour Analgesia, Epidural Anaesthesia; Duration of Labour; Labor, Induced
Keywords: neuraxil analgesia; induced labour
MeSH Terms: interventions — Analgesia, Epidural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- women undergoing labour induction
  Interventions: Procedure: Epidural analgesia for labour pain

INTERVENTIONS:
Procedure: Epidural analgesia for labour pain — Patients were divided into two groups according to repertorised cervical dilatation at the start of analgesia: Group A < 4 centimetres (latent stage according to National Institute for Health and Care Excellence guidelines) and Group B between 4 and 6 centimetres.

SUMMARY:
The aim of this observational study is to assess the effect of early labour analgesia on obstetric and neonatal outcomes in induced labour in primiparous women with a full-term pregnancy whose labour was induced with a Cook balloon or prostaglandins.

It aims to answer whether early labour analgesia (< 4 centimetres of cervical dilation) prolongs the duration of labour. Secondary outcomes will be Incidence of caesarean section, use of oxytocin, onset of fetal heart rate abnormalities within 30 minutes of augmentation, incidence of episiotomy, amount of blood loss, need for epidural catheter repositioning due to inadequate analgesia, onset of breakthrough pain defined as need for "rescue" top-ups within 60 minutes of previous top-ups, Apgar score (at 1 and 5 minutes), neonatal umbilical pH and neonatal intensive care unit admission. Patients who received early partoanalgesia were compared for the proposed outcomes with patients who received partoanalgesia in active labour (cervical dilation > 4 centimetres).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* Primipara;
* Single pregnancy;
* Gestational age > 36 weeks;
* Induced labour with Bishop Score < 6;
* Cervical dilatation at start of analgesia ≤ 6 cm;
* ASA Class 2.

Exclusion Criteria:

* Endouterine fetal death;
* Anhydramnios:
* Trial labour after caesarean section;
* Cardiotocogram class ≥2 before start of analgesia;
* Third trimester bleeding;
* Patient refusal;
* Inability to understand informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnancy
Study Population: women with induced labour undergoing epidual analgesia
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2022-10-21 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Duration of labour | Perioperative/Periprocedural. The investigator traces the information examining the medical chart in a time frame from one day after birth until 6 month from study termination.
  The primary objective is to compare the duration of the first stage of labour (measured in minutes) between women who received early neuraxial analgesia in the latent phase of the first stage and those who received it in the active stage. First stage duration is the time elapsed from the onset of labour, as diagnosed by an experienced obstetrician, until 10 centimetres of cervical dilation is reached.
  The co-primary objective is to compare the duration of the second stage (measured in minutes) between the two populations.
  Second stage duration is the time from 10 centimetres of cervical dilation to birth.
  Data on these outcomes are recorded by the obstetric team in the patient's chart during labour.

SECONDARY OUTCOMES:
Incidence of operative deliveries | Perioperative/Periprocedural. The investigator traces the information examining the medical chart in a time frame from one day after birth until 6 month from study termination.
  The incidence of operative deliveries by obstetrical suction cup for lack of progression of the presented part or presence of fetal heartbeat abnormalities was assessed. Data relating to the mode of delivery and events are recorded in the patient's medical chart by the obstetric team during labour.
Incidence of Episiotomy | Perioperative/Periprocedural. The investigator traces the information examining the medical chart in a time frame from one day after birth until 6 month from study termination.
  The incidence of episitomy due to lack of progression of the presented part or presence of fetal heartbeat abnormalities was assessed. Data on this outcome is recorded in the patient's medical chart by the obstetric team during labour.
Incidence of caesarean section during labour | Perioperative/Periprocedural. The investigator traces the information examining the medical chart in a time frame from one day after birth until 6 month from study termination.
  The incidence of caesarean section in labour was assessed. The causes of caesarean section considered were: first stage prolongation, second stage prolongation, fetal heartbeat abnormalities.Data on this outcome is recorded by the obstetric team in the patient's chart during labour.
Incidence of Obstetric lacerations | Perioperative/Periprocedural. The investigator traces the information examining the medical chart in a time frame from one day after birth until 6 month from study termination.
  The incidence of grade I, II, III obstetric lacerations was evaluated. Data on this outcome is recorded by the obstetric team in the patient's chart during labour.
Oxytocin consumption | Perioperative/Periprocedural. The investigator traces the information examining the medical chart in a time frame from one day after birth until 6 month from study termination.
  The amount of oxytocin used during labour was assessed. Data on this outcome is recorded by the obstetric team in the patient's chart during labour.
  The amount was measured in units per minute.
Peridural catheter repositioning | Perioperative/Periprocedural. The investigator traces the information examining the medical chart in a time frame from one day after birth until 6 month from study termination.
  The incidence of epidural catheter repositioning for inadequate analgesia was measured.
  Analgesia was defined as inadequate if the Visual Analogue Scale > 4 30 minutes after analgesia was administered.
  During labour analgesia, this event was recorded by the anaesthetist on duty in the anaesthesia chart.
Fetal heart rate abnormalities | Perioperative/Periprocedural. The investigator traces the information examining the medical chart in a time frame from one day after birth until 6 month from study termination.
  Fetal heart rate abnormalities occurring within 30 minutes of local anaesthetic or neuroaxial opioid administration have been recorded. The American Congress of Obstetricians and Gynecologists classification was used for the identification of trace abnormalities. Abnormal foetal heart rate are recorded as they occur by the obstetrician in patient's medical chart.
Apgar score | Perioperative/Periprocedural.The investigator traces the information examining the medical chart in a time frame from one day after birth until 6 month from study termination.
  The Apgar score is assessed by a paediatrician using a scale from 0 to 10 at 1 minute and 5 minutes after birth. The information is then recorded in the baby's and mother's medical records.
pH Neonatal umbilical cord | Perioperative/Periprocedural. The investigator traces the information examining the medical chart in a time frame from one day after birth until 6 month from study termination.
  The arterial pH of the umbilical cord is assessed.After delivery the obstetrician takes a sample of umbilical arterial blood to measure pH. The information is then recorded on baby's and mother's medical chart.
Admission to neonatal intensive care unit | Perioperative/Periprocedural.The investigator traces the information examining the medical chart in a time frame from one day after birth until 6 month from study termination.
  This outcome is assessed from the moment of birth until 2 hours after delivery. The event is recorded in the mother's medical record.
Administering a 'rescue' epidural analgesia | Perioperative/Periprocedural.The investigator traces the information examining the medical chart in a time frame from one day after birth until 6 month from study termination.
  The need for a 'rescue' epidural was assessed. The time of administration of each epidural top up was recorded both on patient medical chart and on anaesthesia medical chart. When, after initial benefit, the patient experienced a recurrence of pain (Visual analogue Score greater than four) and needed an additional top up within 60 minutes from previous epidural bolus, the event was registered.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, SC AR3 - Anestesia e Terapia Intensiva Postchirurgica, Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Simpson KR. Cervical Ripening and Labor Induction and Augmentation, 5th Edition. Nurs Womens Health. 2020 Aug;24(4):S1-S41. doi: 10.1016/j.nwh.2020.04.005. PMID 32778395
- [Background] Wong CA, McCarthy RJ, Sullivan JT, Scavone BM, Gerber SE, Yaghmour EA. Early compared with late neuraxial analgesia in nulliparous labor induction: a randomized controlled trial. Obstet Gynecol. 2009 May;113(5):1066-1074. doi: 10.1097/AOG.0b013e3181a1a9a8. PMID 19384122
- [Background] Ohel G, Gonen R, Vaida S, Barak S, Gaitini L. Early versus late initiation of epidural analgesia in labor: does it increase the risk of cesarean section? A randomized trial. Am J Obstet Gynecol. 2006 Mar;194(3):600-5. doi: 10.1016/j.ajog.2005.10.821. PMID 16522386
- [Background] Sng BL, Sia ATH. Maintenance of epidural labour analgesia: The old, the new and the future. Best Pract Res Clin Anaesthesiol. 2017 Mar;31(1):15-22. doi: 10.1016/j.bpa.2017.01.002. Epub 2017 Jan 12. PMID 28625301